CLINICAL TRIAL: NCT02906800
Title: Potentiation of Cisplatin-based Chemotherapy by Digoxin in Advanced Unresectable Head and Neck Cancer Patients
Acronym: DIGHANC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cancer Research and Personalized Medicine (Carpem) (Unknown); Laboratoire d'excellence en immuno-oncologie (Labex) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150401; 2015-003076-78 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-09-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Head and Neck Cancer
Keywords: cisplatin; head and neck cancer; digoxin
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DIGHANC (Experimental): Patients meeting all inclusion /exclusion criteria, will be given 3 cycles of the following regimen: 1) digoxin (0.25 mg/day) for a 7-day period (digitalization time) from Day 1 to Day 7; 2) chemotherapy regimen TPF protocol from Day 8 to D12 (continuous perfusion of fluorouracil for 120h, Cisplatin at Day 10 and Docetaxel at Day 11) administered in combination with digoxin 0.25 mg/day from Day 8 to Day 9; 3) a 15-day period off treatment.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — The digoxin dose will be adjusted to achieve a plasma concentration of 0.6-1.2 ng/ml according to current recommendations in heart failure patients (doses adapted to renal function, comorbidities, concomitant medications, age, and plasma concentration). The risk related to digoxin treatment will be minimized in our study since the duration of exposure to digoxin will be limited to 9 days every 3 weeks for 3 cycles (total duration of treatment 27 days).
  Other Names: Digoxine

SUMMARY:
Introduction: Patients with primary unresectable advanced head and neck squamous cell carcinomas (HNSCC) have a poor prognosis with a median survival of 22 months (Hauswald H Radiat Oncol 2011). They are usually treated with induction chemotherapy followed by radiochemotherapy or platinum-based concomitant radiochemotherapy. Most patients achieve an objective clinical response contrasting with a high rate of local recurrence and distant metastases in the year following radiochemotherapy (Argiris A Ann Oncol 2011). Improvement of the efficacy of chemotherapy remains therefore a major clinical goal for this group of patients. During the past years, the investigators demonstrated that some conventional chemotherapeutics (anthracycline, oxaliplatin…) induce a type of "immunogenic" cell death (ICD) characterized by the exposure of calreticulin on the tumor cell surface, the secretion of ATP and the release of high-mobility group box 1 (HMGB1) resulting in activation of tumor immunity (Galluzzi L Nat Rev Drug Discov 2012). The investigators recently showed that the Na/K-ATPase inhibitor, digoxin, favors ICD, when combined with cisplatin, a drug known not to induce ICD. In preclinical models, a synergy between cisplatin and digoxin which led to a significant therapeutic improvement (Menger L Sci Transl Med 2012) has been observed. This effect seems to be mediated by the immune system as the combined therapy induced intratumor T cell infiltration producing cytokines (Menger L Sci Transl Med 2012).

Hypothesis: Based on our preclinical data, the hypothesis is that adding digoxin to the conventional cisplatin based induction chemotherapy regimen in unresectable advanced HNSCC will increase the efficacy of this therapy via the induction of anti-tumor immunity.

Objectives:

Main: the primary objective is to assess the clinical and biological safety of the combination of digoxin to cisplatin-based chemotherapy.

Secondary: The secondary objectives are to investigate biological markers of efficacy by analyzing the recruitment of functional T cells in tumour biopsies after treatment with the combination of digoxin and chemotherapy.

DETAILED DESCRIPTION:
Introduction:

Patients with primary unresectable advanced head and neck squamous cell carcinomas (HNSCC) have a poor prognosis with a median survival of 22 months (Hauswald H Radiat Oncol 2011). They are usually treated with induction chemotherapy followed by radiochemotherapy or platinum-based concomitant radiochemotherapy. Most patients achieve an objective clinical response contrasting with a high rate of local recurrence and distant metastases in the year following radiochemotherapy (Argiris A Ann Oncol 2011). Improvement of the efficacy of chemotherapy remains therefore a major clinical goal for this group of patients. During the past years, it was demonstrate that some conventional chemotherapeutics (anthracycline, oxaliplatin…) induce a type of "immunogenic" cell death (ICD) characterized by the exposure of calreticulin on the tumor cell surface, the secretion of ATP and the release of HMGB1 resulting in activation of tumor immunity (Galluzzi L Nat Rev Drug Discov 2012). The Na/K-ATPase inhibitor, digoxin, favors ICD, when combined with cisplatin, a drug known not to induce ICD. In preclinical models, a synergy was observed between cisplatin and digoxin which led to a significant therapeutic improvement (Menger L Sci Transl Med 2012). This effect seems to be mediated by the immune system as the combined therapy induced intratumor T cell infiltration producing cytokines (Menger L Sci Transl Med 2012).

Hypothesis:

Based on our preclinical data, the hypothesis is that adding digoxin to the conventional cisplatin based induction chemotherapy regimen in unresectable advanced HNSCC will increase the efficacy of this therapy via the induction of anti-tumor immunity.

Objectives:

Main: the primary objective is to assess the clinical and biological safety of the combination of digoxin to cisplatin-based chemotherapy.

Secondary: The secondary objectives are to investigate biological markers of efficacy by analyzing the recruitment of functional T cells in tumour biopsies after treatment with the combination of digoxin and chemotherapy.

Endpoints:

Primary: grade 3 or 4 clinical or biological toxicity (Adverse Events graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.0)

Secondary:

* Clinical/radiological efficacy monitored after 3 cycles of chemotherapy as assessed by Positron Emission Tomography-Scan (PET-Scan), Magnetic Resonance Imaging (MRI), (computerized tomography-Scan) CT-scan
* Progression Free Survival (PFS) (months)
* Biological efficacy monitored by:

  1. Analysis of the T cells recruitment in biopsies from HNSCC patients after therapy. The T cell recruitment will be considered as significant if T cells increase of at least 25% in post-therapeutic compared to pre-therapeutic biopsies.
  2. Analysis of subpopulations of T cells (CD8+T cells, regulatory T cells (CD4+CD25+Foxp3+ and gamma-delta T cells) in tumor biopsies by immunofluorescence analysis to show a potential higher ratio of effector/regulatory T cells after therapy as previously described (Badoual C et al Clin Cancer Res 2006).
  3. Expression of IFN and IL-17 assessed by quantitative RT-PCR assay (Taq Man) to look for a production of Interferon gamma (IFNgamma) by CD4+ and CD8+T cells and the presence of T cells producing IL-17 as observed in preclinical models, (Menger L Sci Transl Med 2012).

Methodology: Pilot, single arm, open label, phase I/II study.

Study conduct:

Patients meeting all inclusion /exclusion criteria, will be given 3 cycles of the following regimen: 1) digoxin (0.25 mg/day) for a 7-day period (digitalization time) from Day 1 to Day 7; 2) chemotherapy regimen TPF (Taxoter, Platin, 5-FU) protocol from Day 8 to D12 (continuous perfusion of fluorouracil for 120h, Cisplatin at Day 10 and Docetaxel at Day 11) administered in combination with digoxin 0.25 mg/day from Day 8 to Day 9; 3) a 15-day period off treatment.

The digoxin dose will be adjusted to achieve a plasma concentration of 0.6-1.2 ng/ml according to current recommendations in heart failure patients (doses adapted to renal function, comorbidities, concomitant medications, age, and plasma concentration). The risk related to digoxin treatment will be minimized in our study since the duration of exposure to digoxin will be limited to 9 days every 3 weeks for 3 cycles (total duration of treatment 27 days).

Biopsies will be performed before the first digoxin administration and at the end of the 3rd cycle.

Patients with unacceptable adverse events (e.g. patients with grade 3 or 4 toxicities not improving to < grade 1 despite drug hold for 2 weeks) will be withdrawn of the study.

Patients with estimated glomerular filtration rate (estimated by the MDRD formula) decreasing below 60 ml/min/1.73m2 at any time after the TPF chemotherapy during the study will be withdrawn of the study.

Patients will be managed jointly by an oncologist and a cardiologist at the Clinical Investigation Center or at the Oncology and safety and tolerability assessed at each cycle by:

Physical examination including neurological and hearing testing, body weight, WHO performance status Cardiac status: echocardiogram at baseline and daily ECG at rest during each cycle of chemotherapy (from Day 8 to Day 12) and at Day 1 of each cycle and at inclusion.

Plasma digoxin concentration and plasma electrolytes and creatinine (at inclusion, at day 1 at cycles 2 and 3 and everyday during the TPF chemotherapy regimen of each cycle of chemotherapy).

Regular reporting of adverse events (AEs) graded by NCI CTC version 4.0.

An Independent Safety Committee will receive information at the end of the treatment period of each patient, and if a serious adverse event (SAE) occurs. A formal meeting will be held every 3 patients.

Randomisation: none

Duration of participation for each patient: 18 weeks including the inclusion protocol

Length of the study: 28 months 1/2

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, with primary unresectable, advanced (stage III-IV) HNSCC to be treated by cisplatin-based chemotherapy.
* Life expectancy > 12 months.
* Age > 18 and < 70
* WHO PS : 0-2
* Signed informed consent
* creatinine clearance : MDRD > 60ml/min/1,73m2
* Affiliation to the French Social Security Health Care plan

Exclusion Criteria:

* Difficulties planned for the 6 month follow up during the study period
* Swallowing disorder preventing digoxin treatment
* Severe aortic stenosis or idiopathic hypertrophic subaortic stenosis at the pretreatment echocardiography.
* Hypertrophic or dilated or restrictive cardiomyopathy at the pretreatment echocardiography
* Severe cardiac condition contraindicating the use of digoxin (Constrictive pericarditis, acute cor pulmonale, myocarditis…)
* Acute Myocardial infarction within the past 3 months
* Severe ventricular arrhythmias on ECG at rest including frequent ventricular extrasystoles, ventricular tachycardia/fibrillation
* Second and third degree atrio-ventricular block or sick sinus syndrome on resting ECG without pacemaker
* Wolf Parkinson White syndrome on ECG at rest
* Renal insufficiency (estimated glomerular filtration rate by the MDRD formula < 60 ml/min/1.73m2)
* Liver insufficiency (Child-Pugh grades B and C)
* Severe uncorrected electrolyte disturbances (hypercalcemia, hypokaliemia, hypomagnesemia…)
* Known hypersensitivity reaction to digoxin
* Compelling indication for continuous use of digoxin
* Use of drugs contraindicated with oral digoxin (Midodrine, calcium salt, millepertuis, sultopride, phenytoin, yellow fever vaccine, live attenuated vaccine)
* Absence of effective contraception methods for men and women during the study and 6 months after the end of the study
* Pregnancy and breastfeeding at inclusion, during the study and 6 months after the end of the study
* HPV positive tumors (These tumors are associated with very good response to chemotherapy alone)
* History of another cancer which treatment is ongoing

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Appearance of the grade 3 or 4 (Adverse Events graded by NCI CTC version 4.0) clinical or biological toxicity of the combination of digoxin to cisplatin-based chemotherapy during the study | 18 weeks

SECONDARY OUTCOMES:
Clinical response after chemotherapy by fibroscopy (tumor seize) | At 18 weeks
Radiological response after chemotherapy | At 18 weeks
  Measured by TDM, MRI and TEP-Scan (tumor seize, criteria RECIST (Response Evaluation Criteria In Solid Tumours)
Biological efficacy: monitored by analysis of T cells recruitment | At 18 weeks
  Analysis of the T cells recruitment in biopsies from HNSCC patients after therapy. The T cell recruitment will be considered as significant if T cells increase of at least 25% in post-therapeutic compared to pre-therapeutic biopsies
Biological efficacy: monitored by analysis of subpopulations of T cells | At 18 weeks
  Analysis of subpopulations of T cells (CD8+T cells, regulatory T cells (CD4+CD25+Foxp3+ and gamma-delta T cells) in tumor biopsies by immunofluorescence analysis to show a potential higher ratio of effector/regulatory T cells after therapy as previously described (Badoual C et al Clin Cancer Res 2006).
Biological efficacy: expression of IFN gamma assessed by quantitative RT-PCR assay | At 18 weeks
Biological efficacy: expression of IL-17 assessed by quantitative RT-PCR assay | At 18 weeks
Progression Free Survival (PFS): Death or recurrence (clinical and/or radiological analysis) | 10 days after each cycle of chemotherapy and two weeks after the end of the third cycle of chemotherapy
  Death or recurrence (clinical and/or radiological analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane HANS, MD, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, Île-de-France Region, France